CLINICAL TRIAL: NCT05264558
Title: Preparing for the Final Phase of Hepatitis C Elimination in Cairns: An Implementation Trial of a Test and Treat Approach to Reach the Final 30%.
Brief Title: Preparing for the Final Phase of Hepatitis C Elimination. Cairns Final 30%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Cairns Hinterland Health Hospital and Health Services (Unknown); The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16112020
Record Dates: First submitted 2022-02-20; First posted 2022-03-03 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; Standard of Care

STUDY DESIGN:
Intervention Model Description: The model will permit all interventions to be explored for their impact on testing and treatment numbers in the HCV care cascade
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Test and treat (Experimental): This group will receive POC HCV viral load testing via a fingerstick using the Xpert HCV Viral load finger stick point of care test (Cepheid) in addition to the standard of care whole blood conventional laboratory based HCV PCR viral load testing. Participants who return a positive POC HCV viral load result will be provided with Epclusa on the same day as result. Follow up management will be determined by results received from standard of care blood. Service level data will be investigated to estimate HCV targeted treatment numbers prior to intervention arms implementation. Service level data will be measured post intervention periods.
  Interventions: Device: Xpert HCV Viral load finger stick point of care test (Cepheid); Drug: Epclusa 400Mg-100Mg Tablet
- General Practitioner Refresher and Clinic in reach (Other): Perform hepatitis C education for GP and clinic staff at primary health services; on hepatitis testing and treatment at a service level will offer the opportunity to tailor education to the requirements of the clinic and staffing needs.Service level data will be investigated to estimate HCV targeted treatment numbers prior to intervention arms implementation. Service level data will be measured post intervention period
  Interventions: Other: Standard of care
- Incentive and Peer intervention in HCV care cascade (Other): Assess the effectiveness in primary health services of engaging people in hepatitis C testing, and retention throughout the care cascade whilst employing innovative techniques including incentives and peer recruitment.Service level data will be investigated to estimate HCV targeted treatment numbers prior to intervention arms implementation. Service level data will be measured post intervention period
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Xpert HCV Viral load finger stick point of care test (Cepheid) — Xpert HCV VL Fingerstick is an in vitro reverse transcription polymerase chain reaction (RT-PCR) assay for the detection and quantification of Hepatitis C Virus (HCV) RNA in human venous and capillary fingerstick EDTA whole blood. Appropriate pre and post testing counselling will be provided to participants.
  Arms: Test and treat
Drug: Epclusa 400Mg-100Mg Tablet — Same day HCV test and treatment
  Arms: Test and treat
Other: Standard of care — Clinical services will receive additional education and have the option of providing incentives to attendees of service.
  Arms: General Practitioner Refresher and Clinic in reach; Incentive and Peer intervention in HCV care cascade

SUMMARY:
The study aims to assess the impact of models of HCV care on HCV testing, treatment uptake and cure within Cairns. Point of care testing for HCV , with test and treat strategies will be offered within a primary care service.

DETAILED DESCRIPTION:
Available testing and treatment data will be explored pre and post the intervention period of the project within Cairns Hinterland health services that provide hepatitis C care.

Test and treat strategies of the project will include:

Part A: Same day test and treat clinical trial. The study will explore a 'same day test and treat' model to determine the impact on HCV treatment initiation and cure within a primary care service that recognises that they see people at risk of hepatitis C that are transient, and struggle to return to a care provider to engage in hepatitis C testing and care.

1. HCV RNA point of care (POC) testing
2. Epclusa (Sofosbuvir/Velpatasvir 400mg/100mg) course initiated at same day of visit following a +ve HCV RNA result from the POC test.

Part B: Refresher and clinic in reach support work Primary care service/ General practitioner education and training ~1 hour in-person training for all clinic staff on hepatitis C testing, treatment, retention in HCV care cascade.

Part C: Services evaluation with incentive and peer intervention in HCV care cascade.

ELIGIBILITY:
Inclusion Criteria:

* attending primary health care service of CHHS aged 18 years or over

Exclusion Criteria: only for intervention arm test and treat

* Known to have hepatitis B or HIV infection
* Known to have cirrhosis
* Previous treatment with direct acting antivirals
* Previously received interferon-based hepatitis C treatment that did not work
* Women that are pregnant or breastfeeding
* Already receiving hepatitis C treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
HCV testing | 12 months
  The number of participants who receive HCV testing in each of the arms
HCV treatment | 12 months
  The number of participants who start HCV treatment in each of the arms

CONTACTS AND LOCATIONS:
Locations (1):
- Cairns and Hinterland Hospital and Health Service, Cairns, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No